CLINICAL TRIAL: NCT05415267
Title: Comparison of Immunity-boosting Regimens for COVID-19 Upon Initiation of Immunosuppressive Therapy
Brief Title: Immunosuppression and COVID-19 Boosters
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Seqirus Pty Ltd, Australia (Unknown); Medical Research Future Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIRCUIT Study
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: Vaccination; Immunology
MeSH Terms: conditions — COVID-19 | interventions — Tetanus Toxoid; Vaccines; COVID-19 Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 Arm A (Active Comparator): Immediate SARS-CoV-2 booster at week 0 and booster of combined diphtheria toxoid/tetanus toxoid (dT vaccine) at week 24.
  Interventions: Biological: diphtheria and tetanus toxoids (adsorbed) vaccine; Biological: COVID-19 vaccine
- Group 1 Arm B (Active Comparator): dT vaccine at week 0 and SARS-CoV-2 deferred booster at week 24.
  Interventions: Biological: diphtheria and tetanus toxoids (adsorbed) vaccine; Biological: COVID-19 vaccine
- Group 2 Arm C (Active Comparator): Immediate SARS-CoV-2 booster at week 0.
  Interventions: Biological: COVID-19 vaccine
- Group 2 Arm D (Active Comparator): Delayed SARS-CoV-2 booster at week 24
  Interventions: Biological: COVID-19 vaccine

INTERVENTIONS:
Biological: diphtheria and tetanus toxoids (adsorbed) vaccine — The diphtheria/tetanus toxoids vaccine will be given to participants enrolled into Group 1 as a comparator vaccine to the mRNA COVID-19 booster vaccine with the aim of determining whether the results related to COVID-19 vaccine timing also apply to more traditional protein-based vaccines.
  Other Names: ADT Booster
  Arms: Group 1 Arm A; Group 1 Arm B
Biological: COVID-19 vaccine — All participants will receive a COVID-19 booster vaccination at either week 0 or week 24 depending on their randomised study arm

SUMMARY:
It is important people receiving immunosuppressive therapy are provided with the best protection against COVID-19 because they are at greater risk of severe illness should they become infected. As severe immunosuppression can reduce the efficacy of COVID-19 vaccination, doctors agree that COVID-19 boosters is are important to maximise the vaccine response in these people. However, we don't currently know the best time to give booster vaccines to people about to start immunosuppressive therapy. This research aims to address this knowledge gap by examining whether the greatest protection is provided by giving the COVID-19 booster just before the immunosuppressive therapy starts or by waiting and giving the booster 6 months after treatment start. At the 6-month timepoint, in many cases the more intensive immunosuppression is often weaning and the immune system is starting to rebuild.

DETAILED DESCRIPTION:
Current guidelines for SARS-CoV2 vaccination in immunosuppressed populations are based on limited evidence. Additionally, guidelines for the use of SARS-CoV2 vaccines in autoimmune populations are somewhat contradictory, with the 2019 European League Against Rheumatism (EULAR) recommendations including advice to where possible administer booster vaccinations prior to commencing immunosuppression but to preferably vaccinate while the autoimmune disease is not active. In haematological conditions it is suggested that vaccination occur prior to B cell depletion therapies e.g. rituximab, or >6 months after its use. While these guidelines were developed for non-live vaccines in general, the evidence for COVID-19 vaccines is almost entirely based on expert opinion. Clearly, with these gaps and inconsistencies in the clinical guidelines there is equipoise for the optimal timing of a booster vaccination. One of the difficulties in this field is the wide diversity of patients receiving a variety of immunosuppressive therapies. We have therefore taken a pragmatic 'real-world' approach in our design by focusing on two broad patient groups that are more specifically stratify based on pre-define disease conditions and specific treatments.

Recent data studying COVID-19 vaccine responses in patients on immunosuppressive therapies for autoimmune/inflammatory conditions demonstrate the greatest compromise in anti-Spike IgG occurs in those receiving combination immunosuppression particularly regimens that include methotrexate and other antimetabolites, and B cell depleting therapies. In patients with haematological malignancies the lowest vaccine responses were seen in chronic lymphocytic leukaemia, lymphoma and multiple myeloma. In patients with a haematological malignancy who have undergone a bone marrow transplant, immunisation to COVID-19 <6 months following transplantation resulted in poor IgG response to vaccine, while those immunised >6 months post-transplant had superior responses. In contrast, other targeted therapies including the integrin inhibitor vedoluzimab or anti IL-17/23 therapy (in the absence of concurrent methotrexate) have relatively preserved response to the initial vaccine regimen. Given the available data, we propose to study defined populations of two major immunosuppressed patient groups: Group 1): Haematological Malignancy (excluding bone marrow transplant recipients) and Autoimmune/Inflammatory Disease, and Group 2: Autologous and Allogeneic Bone marrow transplant (BMT) recipients. We will compare the difference between an immediate COVID-19 "booster" dose and a deferred COVID-19 "booster". In Group 1 "Immediate" is defined as prior to the commencement of moderate-to-severe immunosuppression and "Deferred" is defined as 6 months post commencement of moderate-to-severe immunosuppression. For Group 2 BMT patients, current national guidelines recommend 3 doses of pre-BMT COVID-19 vaccines followed by 3 doses of post-BMT COVID-19 vaccines initiated 6 months post-BMT. In Group 2 "Immediate" is defined as 6 months post-BMT and "Deferred" as >12 months post-BMT.

The primary endpoint will be the integrated area under the curve (AUC) of anti-SARS-CoV-2 neutralizing antibody (NAb) activity over the first year of immunosuppression. At present the level of anti-SARS-CoV-2 is the most robust correlate of protection against COVID-19. In both study Groups the comparator of a delayed boost at 6 months is based on the premise of maximising peak NAb responses by administering the booster after induction therapy is completed. Such a delay must be weighed against the risk of reduced immunity and breakthrough COVID-19 infection during this period. Such a risk will be monitored closely during the study with scheduled interim safety analyses and reviews by an independent data safety monitoring board (DSMB).

Participants in Group 1 will also receive a single diphtheria/tetanus (dT) toxoid booster as a comparator vaccine with the aim of determining whether the results of the optimal timing of the COVID-19 booster also apply to more traditional protein vaccines. If this is found to be the case, the results of this study may have broader implications for the vaccinology field and optimal clinical guidelines.

Primary Objective: to determine the anti-SARS-CoV-2 NAb response over 12 months from a booster with a SARS-CoV2 vaccine over 12 months in a population who; Group 1: are commencing moderate-to-severe immunosuppression for treatment of either a haematological malignancy (excluding BMT patients) or an autoimmune/inflammatory condition and are previously fully-immunised (i.e. had received 3 or more doses of a SARS-CoV-2 vaccine including combinations) or, Group 2: have recently undergone a bone marrow transplant for a haematological malignancy and have previously received 3 post-BMT doses of a SARS-CoV-2 vaccine including combinations.

We will determine the difference between the booster being administered as follows: Group 1: immediately prior to starting moderate-to-severe immunosuppression or at 6 months after therapy start, by monitoring the relative sustained immunogenicity over 1 year. Group 2: immediately at 6-months post-BMT or deferred until >12 months post-BMT.

Secondary Objectives:

1. To assess a range of secondary immunological endpoints including:

   1. . To quantitate antibodies to tetanus toxoid integrated over the 12-month period post-randomisation.
   2. . To assess the safety and efficacy of the two approaches (immediate or deferred vaccination) including any indication of vaccine-induced disease flares and any breakthrough infections with SARS-CoV-2.
   3. . To analyse the response to the SARS-CoV2 vaccine including: i. Breadth of NAb against the SARS-CoV-2 variants of concern (VOC) ii. The kinetics of neutralizing antibody over time including responses to VOC iii. Memory T cell, B cell and natural killer (NK) cell responses to peptide sets representing different domains of the SARS-CoV-2 spike protein
2. To assess these responses in populations stratified by broad disease type (i.e. haematological malignancy (excluding bone marrow transplant recipients), autoimmune/inflammatory disease or haematological malignancy post-BMT and different modes of immunosuppression e.g. chemotherapy, bone-marrow transplant, B-cell depleting therapies, cytokine inhibition.
3. To use a computational biology approach to a) model the level of protection over time based on neutralizing antibody levels and b) model the boosting and decay of anti-Spike IgG, specific memory B, T and NK cell response to provide information on the impact of immunosuppression on vaccine protection over time.
4. To use this evidence-base to inform policies regarding timing of additional SARS-CoV-2 boosters in vulnerable populations about to commence immunosuppression/or following bone marrow transplant. These findings will identify those patient groups most appropriate for synthetic COVID-19 monoclonal antibodies and will contribute to our understanding of vaccinology in the setting of immunosuppression and BMT more broadly, an area that remains poorly understood.
5. To compare the change in health-related quality of life over time between "immediate" and "deferred" booster strategies.

Participant population

Participants will be recruited through a clinical network of specialist physicians at Sydney hospitals who will be recruiting from their Departments of Haematology, Immunology, Rheumatology, Gastroenterology and Neurology. A total of 320 participants will be enrolled into one of two Groups will be enrolled as outlined below:

Group 1: will comprise 280 participants commencing immunosuppression for the management of a pre-defined group of haematological malignancies (excluding bone marrow transplant recipients) or autoimmune/inflammatory conditions as outlined below Group 2: will comprise 40 participants who have undergone a bone marrow transplant for a haematological malignancy as outlined below.

Group 1:

Haemato-Oncology: Haematological Malignancy (excluding bone marrow transplant recipients) - B-CLL; Follicular or Marginal Zone Lymphoma; Multiple Myeloma; Diffuse large B-cell lymphoma

Systematic Autoimmunity: to include: ANCA associated-vasculitis; polyarteritis nodosa; Churg-Strauss syndrome; ankylosing spondylitis; autoimmune hepatitis; IgG4 disease; inflammatory bowel disease; psoriatic arthritis; psoriasis; rheumatoid arthritis; systemic lupus erythematosus; Sjogren's syndrome; myasthenia gravis; and multiple sclerosis. Receiving the following agents:

B-Cell Depletion therapies e.g. rituximab, ocrelizumab, ofatumumab (N=40) Anti-metabolite therapies: azathioprine, calcineurin inhibitors, mycophenolate or methotrexate (Moderate Immunosuppression) (N=40) Tumour necrosis factor alpha inhibition (N=40) (with or without azathioprine or methotrexate or leflunomide to prevent anti-drug antibodies) Cyclophosphamide or alemtuzumab (severe immunosuppression) (N=40) Janus Kinase (JAK) inhibitors +/- leflunomide (N=40) Anti-IL-17 and/or 23 monoclonal antibodies e.g. sekukinumab (N=40).

Group 2:

Bone Marrow Transplant (N=40) Haematological malignancy - autologous or allogenic-transplant (excluding for treatment of a primary Immunodeficiency).

Study Design

This is a randomised, open-label, multi-centre clinical trial to be conducted over 52 weeks.

Participants will be enrolled into one of two Groups as described above. Group 1 participants will be screened to confirm their diagnosis and that they are to commence treatment that involves >1 year on moderate-to-severe immunosuppressive therapy. Participants will be randomised in a 1:1 ratio to either Arm A; Immediate SARS-CoV-2 booster at week 0 and a booster of combined diphtheria toxoid/tetanus toxoid (dT vaccine) at 24 weeks, or Arm B; dT vaccine at week 0 and a deferred SARS-CoV-2 booster at 24 weeks. Participants will be followed until week48 and attend study visits at screening, randomisation, vaccination* and then at weeks 1, 4, 12, 24, 25, 28, 36 and 48.

Group 2 participants will be screened and randomised in a 1:1 ratio to either Arm C; Immediate SARS-CoV-2 booster at week 0 or Arm D delayed SARS-CoV-2 booster at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged at least 18 years
* Previously vaccinated with 2 (or more) doses of any licensed COVID-19 vaccine who requires initiation of moderate-to-severe immunosuppression; most recent COVID-19 vaccine dose must have been given > 3 months prior
* Planned significant immunosuppressive therapy for at least 1 year
* No cyclophosphamide, alemtuzumab or rituximab treatment in the past 5 years. Note: patient may have concurrent steroids with any treatments listed in protocol
* Voluntarily given written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Has underlying primary immunodeficiency
* Has received or likely to receive intravenous/subcutaneous immunoglobulin (IVIg/ScIg).
* Projected treatment is likely to involve plasma exchange
* Contraindication to receipt of SARS-CoV-2 vaccine
* Intolerance of or previous allergic reaction to tetanus vaccination
* Patients switching immunosuppressive therapies following enrolment with an absolute lymphocyte count <0.5 x 109/L immediately prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
anti-SARS-CoV-2 neutralising antibody (NAb) response over 12 months | 48 weeks
  Integrated time-weighted area under the curve (AUC) change from baseline in anti-SARS- CoV-2 NAb over 12 months from a SARS-CoV-2 vaccination

SECONDARY OUTCOMES:
Tetanus toxoid NAb response over 12 months | 48 weeks
  Integrated time-weighted AUC change from baseline in tetanus toxoid NAb over 12 months from a diphtheria/tetanus toxoids vaccination
Safety of immediate versus deferred COV-19 booster vaccination | 48 weeks
  Comparison of adverse events and disease flares between immediate and deferred arms in Group 1 and Group 2
Efficacy of immediate versus deferred COV-19 booster vaccination | 48 weeks
  Comparison of COVID-19 disease flares between immediate and deferred arms in Group 1 and Group 2

CONTACTS AND LOCATIONS:
Overall Officials: Sarah C Sasson, PhD, Principal Investigator — The Kirby Institute UNSW Sydney
Locations (5):
- Australia (5):
  - Blacktown Hospital, Blacktown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord General Repatriation Hospital, Concord, New South Wales
  - St Vincent's Hospital, Sydney, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zorger AM, Hirsch C, Baumann M, Feldmann M, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with haematological malignancies. Cochrane Database Syst Rev. 2025 May 21;5(5):CD015530. doi: 10.1002/14651858.CD015530.pub2. PMID 40396505